CLINICAL TRIAL: NCT02879981
Title: A Pilot, Multicentric and Observational Study of Safety of Sulfamethoxazole + Trimethoprim + Guaifenesin (Balsamic Bactrim) in Pediatric Patients With Acute Bronchitis
Brief Title: A Safety Study of Balsamic Bactrim in Pediatric Participants With Acute Bronchitis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30017
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — Guaifenesin; Sulfamethoxazole; Trimethoprim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pediatric Participants With Acute Bronchitis: Pediatric participants receiving treatment for acute bronchitis with Balsamic Bactrim according to standard of care and in line with the current summary of product characteristics (SPC) / local labeling and who have no contraindication to Balsamic Bactrim as per the local label will be observed for safety.
  Interventions: Drug: Guaifenesin; Drug: Sulfamethoxazole; Drug: Trimethoprim

INTERVENTIONS:
Drug: Guaifenesin — Administration of treatment will be according to treating physician's recommendation under local labeling. The study protocol does not specify any treatment regimen.
Drug: Sulfamethoxazole — Administration of treatment will be according to treating physician's recommendation under local labeling. The study protocol does not specify any treatment regimen.
Drug: Trimethoprim — Administration of treatment will be according to treating physician's recommendation under local labeling. The study protocol does not specify any treatment regimen.

SUMMARY:
This pilot, multicentric and observational study will assess the safety of sulfamethoxazole + trimethoprim + guaifenesin (Balsamic Bactrim) in pediatric participants with acute bronchitis. Administration of treatment will be according to treating physician's recommendation under local labeling.

ELIGIBILITY:
Inclusion Criteria:

* Participants starting treatment with Bactrim Balsamic suspension
* Participants with a clinical diagnosis of acute bronchitis (cough with or without sputum production less than 30 days) according to the medical criteria

Exclusion Criteria:

* Participants who have started treatment with another antibiotic at the time of the visit
* Participants with no respiratory infections
* Participants with mental disorders that do not permit the clinical evaluation of the participant according to the treating physician's criteria
* Participants with severe hepatic parenchymal damage
* Participants with severe renal failure making it difficult to monitor drug plasma concentration
* Participants with hypersensitivity to any of Balsamic Bactrim active ingredients, excipients, and/or sulfas

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric participants receiving treatment for acute bronchitis with Balsamic Bactrim according to standard of care and in line with the current summary of product characteristics (SPC) / local labeling and who have no contraindication to Balsamic Bactrim as per the local label.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events Related to Balsamic Bactrim as Assessed by Treating Physician | From Day 1 up to end of observation (up to 10 days)

SECONDARY OUTCOMES:
Percentage of Participants With Balsamic Bactrim Dose Change (Increase or Decrease) | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Dose Change by Reason for Change | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Change in Balsamic Bactrim Frequency of Administration | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Dose Interruption | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Treatment Discontinuation | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Treatment Reintroduction After Discontinuation | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Compliance to Balsamic Bactrim Treatment According to Local Label, as Assessed by Treating Physician | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Predisposing Factors (Categories) for Safety (No specific predefined factors, these will be decided based on observations during study) | From Day 1 up to end of observation (up to 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Peru (3):
  - Hospital Emergencias Pediatricas; Unidad de Investigación Pediátrica, La Victoria
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Clínica Anglo Americana-CENTRO DE INVESTIGACION PEDIATRIA CAA, San Isidro

REFERENCES:
- [Derived] Falcon M, Iberico C, Guerra F, Reyes I, Felix E, Flores M, de Los Rios J, Diaz ME, Casas A, Sanchez-Gambetta S, Carrasco R. A pilot study of safety of sulfamethoxazole, trimethoprim and guaifenesin in pediatric and adult patients with acute bronchitis. BMC Res Notes. 2019 Mar 4;12(1):119. doi: 10.1186/s13104-019-4150-2. PMID 30832720